CLINICAL TRIAL: NCT06194487
Title: Efficacy Evaluation of Collagen Drink Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23-073-A
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo drink (Placebo Comparator): consume 1 bottle (50mL) per day
  Interventions: Dietary Supplement: Placebo drink
- MAXI Collagen drink (Experimental): consume 1 bottle (50mL) per day
  Interventions: Dietary Supplement: MAXI Collagen drink
- Normal fish collagen drink (Active Comparator): consume 1 bottle (50mL) per day
  Interventions: Dietary Supplement: Normal fish collagen drink

INTERVENTIONS:
Dietary Supplement: Placebo drink — consume 1 bottle (50mL) per day
  Arms: Placebo drink
Dietary Supplement: MAXI Collagen drink — consume 1 bottle (50mL) per day
  Arms: MAXI Collagen drink
Dietary Supplement: Normal fish collagen drink — consume 1 bottle (50mL) per day
  Arms: Normal fish collagen drink

SUMMARY:
To assess MAXI Collagen drink on skin condition improvement

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 35-65 years old

Exclusion Criteria:

* Subject with skin surface damage larger than $50 coin area.
* Subject who had skin allergies caused by diet or undrwent cosmetic or medical treatment within 6 months.
* Subject who is a vegetarian and allergic to seafood, alcohol or listed ingredients in the product.
* Students who are currently taking courses taught by the principal investigator of this trial.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
The change of skin collagen density | Day 0, Day 7, Day 28
  DermaLab® Series SkinLab Combo was utilized to measure skin collagen density. Units: arbitrary units
The change of skin elasticity | Day 0, Day 7, Day 28
  Cutometer® Dual MPA 580 was utilized to measure skin elasticity. Units: arbitrary units
The change of skin moisture | Day 0, Day 7, Day 28
  Corneometer® CM825 was utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120
The change of skin texture | Day 0, Day 7, Day 28
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units

SECONDARY OUTCOMES:
The change of transepidermal water loss (TEWL) | Day 0, Day 7, Day 28
  Tewameter® TM 300 was utilized to measure TEWL. Units: g/hm²
The change of skin wrinkles | Day 0, Day 7, Day 28
  VISIA Complexion Analysis System was utilized to measure skin wrinkles. Units: arbitrary units
The change of skin pores | Day 0, Day 7, Day 28
  VISIA Complexion Analysis System was utilized to measure skin pores. Units: arbitrary units
The change of skin colour | Day 0, Day 7, Day 28
  PANTONE® CAPSURE™ RM200-PT01 was utilized to measure skin colour. Units: arbitrary units
The change of self-assessment skin condition | Day 0, Day 7, Day 28
  A self-assessment questionnaire was collected to evaluate skin condition

OTHER OUTCOMES:
The change of liver function biomarkers (GOT, GPT) of blood | Day 0, Day 28
  Fasting venous blood was sampled to measure liver function biomarkers
The change of renal function biomarkers (creatinine, BUN) of blood | Day 0, Day 28
  Fasting venous blood was sampled to measure renal function biomarkers
The change of fasting blood glucose | Day 0, Day 28
  Fasting venous blood was sampled to measure blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Tzu Fang Hsu, Principal Investigator — Department of Applied Cosmetology, Hungkuang University
Locations (1):
- Department of Applied Cosmetology, Hungkuang University, Taichung, Taiwan